CLINICAL TRIAL: NCT02256293
Title: Acceptability and Feasibility of an ACT-Based Group to Improve Diabetes Self-Management
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00040489
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2014-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Therapy (Experimental): Diabetes self-management group based on Acceptance and Commitment Therapy (ACT).
  Interventions: Behavioral: Diabetes self-management group based on Acceptance and Commitment Therapy (ACT).

INTERVENTIONS:
Behavioral: Diabetes self-management group based on Acceptance and Commitment Therapy (ACT). — The group sessions will be lead by a clinician trained in Acceptance and Commitment Therapy and will meet at Duke Medical Center for 1 ½ hours once a week for a total of 8 weeks. During group sessions, participants will identify how avoidance of difficult thoughts and feelings about diabetes has interfered with diabetes management and learn alternative ways of coping with these experiences. The group sessions are intended to supplement regular medical treatment; thus it is important that subjects continue to have diabetes symptoms monitored by their current treatment provider.

SUMMARY:
Individuals with diabetes often report that difficult thoughts and feelings about diabetes interfere with making healthy choices with regards to diabetes management. The purpose of this study is to evaluate a diabetes self-management group based on Acceptance and Commitment Therapy (ACT). ACT is a new behavior therapy that has been found to be useful in treating psychological and behavioral difficulties. We are interested in whether individuals with diabetes will like an ACT-based diabetes management group and whether they find the group helpful.

DETAILED DESCRIPTION:
The goal of the current study is to assess the acceptability and feasibility of an acceptance-based group to improve diabetes self-management among individuals with Type 1 Diabetes. Interested individuals will participate in a weekly acceptance-based therapy group focusing on improving diabetes management (e.g., adherence to dietary recommendations, appropriate insulin dosing) for a total of 8 weeks. Participants will also be asked to complete questionnaires both pre and post treatment. Questionnaires will assess diabetes management and acceptability of the group (post treatment only). Regular medical monitoring is required for participation in the current study. Participants will be asked to provide consent to contact their current medical provider in order to confirm that the participant's is receiving regular medical monitoring for diabetes care and that providers are aware of their patient's participation in group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnosed with type 1 diabetes
* Currently monitored by a physician for their diabetes

Exclusion Criteria:

* Current or history of psychosis or mania
* Current substance abuse
* Non-English Speaking
* Deficits in intellectual functioning that preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 8 weeks
  Acceptability of treatment as measured by a post-intervention questionnaire.

SECONDARY OUTCOMES:
Diabetes self-management | 8 weeks
  Changes in diabetes self-management as measured by pre and post-intervention questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Merwin, PhD, Principal Investigator — Duke University